CLINICAL TRIAL: NCT03967405
Title: A Prospective Evaluation of Clinical Equivalence Between i:X and PID
Brief Title: A Prospective Evaluation of Clinical Equivalence Between iX and PID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-002
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Wound
Keywords: Wound; Imaging
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MolecuLight PID — Hand-held, real-time fluorescence imaging device

SUMMARY:
Patients with chronic wounds will be imaged using 2 imaging devices. Two types of images will be acquired with each device, a standard photograph (ST-image) and a fluorescence image (FL-image). The images captured with the 2 imaging devices will be compared off-line by many interpreters to assess for any differences in the images that would alter a clinical decision.

DETAILED DESCRIPTION:
Patients (n = 50) with chronic wounds will be imaged using 2 imaging devices. Two types of images will be acquired with each device, as standard photograph (ST-image) and a fluorescence image (FL-image). The images captured with the 2 imaging devices will be compared off-line by many interpreters to assess for any differences in the images that would alter a clinical decision.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects presenting at an advanced outpatient wound care clinic with wound(s) of unknown infection status
2. 18 years of age or older

Exclusion Criteria:

1. Treatment with an investigational drug within 1 month before study enrollment
2. Subjects with recent (<30 days) biopsy or curettage of target wound
3. Subjects with wounds that cannot be completely imaged by study device due to anatomic location
4. Unable or unwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic wounds
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Concordance | 2 months
  The inter-reader concordance of the iX and PID FL-images together is not less than the inter-reader concordance of the iX FL-images alone.

SECONDARY OUTCOMES:
Sensitivity and Specificity | 2 months
  Sensitivity and specificity for detection of moderate/heavy bacterial load of PID FL-images to be equal to or greater than that of i:X FL-images when validated by microbiology gold truth

OTHER OUTCOMES:
Bacterial Load quantification by sampling | 2 months
  Quantify difference in bacterial load reported by sampling using standard Levine technique (swabbing) compared to FL image-guided curettage scraping.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Linden, Principal Investigator — Judy Dan Research and Treatment Center
Locations (1):
- Judy Dan Research and Treatment Center, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to disseminate information to patients. If patients ask for their information then they will be provided a response with the most up to date information.